CLINICAL TRIAL: NCT06890741
Title: Influance of 6000m Ergometer Test on Inflammatory, Permeability Markers and Iron Status.
Brief Title: Inflamation, Gut Leakage, Iron Status After 6000m Ergometer Test in Elite Rowers.
Acronym: 6000m
Status: Completed | Type: Observational
Sponsor: Poznan University of Physical Education (Other)
Responsible Party: Sponsor
Other Study IDs: Rowers6000m 2023
Record Dates: First submitted 2025-03-17; First posted 2025-03-24 (Actual); Last update posted 2025-03-27 (Actual); Status verified 2023-11

CONDITIONS: Endothenial Dysfunction; Iron Status; Oxidative Stress
Keywords: endotoxin; gut permeability; gastrointestinal function; iron status; oxidative stress
MeSH Terms: interventions — Exercise Test

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- elite rowers
  Interventions: Other: exercise test

INTERVENTIONS:
Other: exercise test — Participant perforemed 6000m ergometer test.

SUMMARY:
The influence of a 6000m ergometer test on the markers of gut injury, endotoxemia, iron status, stress and inflammation in elite rowers.

DETAILED DESCRIPTION:
The principal objective of our study was to assess gut permeability after completing a 6000-meter rowing test. The study was performed at the beginning of a competitive training phase. Eighteen elite Polish Rowing Team rowers participated in the study after applying the inclusion/exclusion criteria. The participants performed a 6000-meter ergometer test. Blood samples were taken before the test, after exercise, and after 1 hour of restitution. Parameters, such as I-FABP (intestinal fatty acid binding protein), LPS (lipopolysaccharide), LBP (lipopolysaccharide binding protein), claudin3, ferritin, transferrin, hepcidin, IL-6 (Interleukin-6), HO-1 (Heme Oxygenase 1), and ACSL4 (Long-chain-fatty-acid-CoA ligase 4 ) were determined using appropriate biochemical tests.

ELIGIBILITY:
Inclusion Criteria:

* minimum five years of training,
* five training sessions per week minimum,
* total training time minimum of 240 minutes,
* membership in the Polish Rowing Team,
* finishing the 6000-meter ergometer test.

Exclusion Criteria:

* antibiotic therapy within the last three months,
* probiotics and prebiotics within the last three months,
* dietary regime,
* gastrointestinal diseases.

Ages: 18 Years to 24 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Male rowers age 18 - 24 years.
Sampling Method: Non-Probability Sample
Enrollment: 21 (Actual)
Dates: Start 2023-11-01 (Actual); Primary Completion 2023-11-10 (Actual); Study Completion 2023-11-10 (Actual)

PRIMARY OUTCOMES:
I-FABP (intestinal fatty acid binding protein)to measure epithelial wall injury | Blood samples was taken from the cubital vein at three-time points: before each stress test (after overnight fasting), one minute after the end of the test, and after a 1-hour recovery period
  I-FABP concentration measured in blood [ng/ml] using commercially available enzyme-linked immunosorbent assays
LBP (lipopolysaccharide binding protein) to measure endotoxin | Blood samples was taken from the cubital vein at three-time points: before each stress test (after overnight fasting), one minute after the end of the test, and after a 1-hour recovery period
  LBP concentration measured in blood [ug/ml] using commercially available enzyme-linked immunosorbent assays
Claudin 3 to measure tight junction leakage | Blood samples was taken from the cubital vein at three-time points: before each stress test (after overnight fasting), one minute after the end of the test, and after a 1-hour recovery period
  claudin 3 concentration measured in blood [ng/ml] using commercially available enzyme-linked immunosorbent assays
LPS (lipopolysaccharide) to measure endotoxin | Blood samples was taken from the cubital vein at three-time points: before each stress test (after overnight fasting), one minute after the end of the test, and after a 1-hour recovery period
  LPS concentration measured in blood [EU/Ll] using commercially available enzyme-linked immunosorbent assays
Lactic acid to measure fatigue after the race | Blood samples was taken from earlobe at two-time points: before each stress test (after overnight fasting), one minute after the end of the test.
  Lactate concentration measured in capillary blood from earlobe [mmol/L] using a commercially available kit (Diaglobal, Berlin, Germany)
Ferritin to measure iron status | Blood samples will be taken from the cubital vein at three-time points: before each stress test (after overnight fasting), one minute after the end of the test, and after a 1-hour recovery period.
  Ferritin concentration measured in blood [ng/ml] using commercially available enzyme-linked immunosorbent assays
Transferrin to measure iron status | Blood samples will be taken from the cubital vein at three-time points: before each stress test (after overnight fasting), one minute after the end of the test, and after a 1-hour recovery period.
  Transferrin concentration measured in blood [mg/ml] using commercially available enzyme-linked immunosorbent assays
Hepcidin to measure iron status | Blood samples will be taken from the cubital vein at three-time points: before each stress test (after overnight fasting), one minute after the end of the test, and after a 1-hour recovery period.
  Hepcidin concentration measured in blood [ng/ml] using commercially available enzyme-linked immunosorbent assays
IL-6 (Interleukin-6) to measure inflammation | Blood samples will be taken from the cubital vein at three-time points: before each stress test (after overnight fasting), one minute after the end of the test, and after a 1-hour recovery period.
  IL-6 concentration measured in blood [ng/l] using commercially available enzyme-linked immunosorbent assays.
HO-1 (Heme Oxygenase 1) to measure oxidative stress | Blood samples will be taken from the cubital vein at three-time points: before each stress test (after overnight fasting), one minute after the end of the test, and after a 1-hour recovery period.
  HO-1 concentration measured in blood [ng/ml] using commercially available enzyme-linked immunosorbent assays
ACSL4 (Long-chain-fatty-acid-CoA ligase 4 ) to measure oxidative stress | Blood samples will be taken from the cubital vein at three-time points: before each stress test (after overnight fasting), one minute after the end of the test, and after a 1-hour recovery period.
  ACSL4 concentration measured in blood [pg/ml] using commercially available enzyme-linked immunosorbent assays.

SECONDARY OUTCOMES:
energy | day before test, in the morning before the test
  energy [kcal ]of food intake measured by 24h dietary recall
protein | day before test, in the morning before the test
  protein [g ]of food intake measured by 24h dietary recall
carbohydrate | day before test, in the morning before the test
  carbohydrate [g ]of food intake measured by 24h dietary recall
fat | day before test, in the morning before the test
  fat [g ]of food intake measured by 24h dietary recall
fiber | day before test, in the morning before the test
  fiber [g ]of food intake measured by 24h dietary recall
body mass | in the morning before the test
  Body mass [kg] measured by electronic scale to the nearest 0,05 kg (Tanita BC 418 MA Tanita Corporation, Tokyo, Japan).
Body composition - water | in the morning before the test
  % of body water measured by electronic scale (Tanita BC 418 MA Tanita Corporation, Tokyo, Japan).
Body composition - fat | in the morning before the test
  % of body fat measured by electronic scale (Tanita BC 418 MA Tanita Corporation, Tokyo, Japan).
Lean body mass | in the morning before the test
  Lean body mass [kg] measured by electronic scale to the nearest 0,05 kg (Tanita BC 418 MA Tanita Corporation, Tokyo, Japan).
Height | in the morning before the test
  Prior to the exercise test, we measured the anthropometric parameters, including height (Seca 213 Hamburg, Deutschland) [cm]
Gastrointestinal sypthomps self reported scale | up to 1 hours after the test
  10 point scale were 10 is a outcome of the worst severity

CONTACTS AND LOCATIONS:
Locations (1):
- Poznan University of Physical Education, Gorzów Wielkopolski, Lubusz Voivodeship, Poland

IPD SHARING:
Plan to Share IPD: No